CLINICAL TRIAL: NCT01858012
Title: Impact of Hepatitis C on Insulin Sensitivity and Insulin Secretion in Latinos
Brief Title: Insulin Resistance in HCV Infection
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: UCSF 10-00922
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Insulin Resistance
Keywords: insulin resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum samples and liver tissue specimens for analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HCV infection: patients with hepatitis C infection
  Interventions: Behavioral: Moderate alcohol cessation
- non-HCV infection: healthy controls
  Interventions: Behavioral: Moderate alcohol cessation

INTERVENTIONS:
Behavioral: Moderate alcohol cessation — patients will have moderate alcohol use discontinued for 6 weeks and have before and after alcohol cessation clinical and metabolic assessment and also patients with hepatitis C who have undergo therapy for hepatitis C may have repeat clinical and metabolic assessement
  Other Names: Hepatitis C therapy

SUMMARY:
The study hypothesis is that the means by which HCV induces glucose intolerance is through impairment of B-cell function and compensatory hyperinsulinemia in predisposed Latinos with insulin resistance and that HCV eradication improves these abnormalities. It is also hypothesized that moderate alcohol consumption impact insulin sensitivity and secretion with Latinos with or without HCV infection.

DETAILED DESCRIPTION:
The study hypothesis is that the means by which HCV induces glucose intolerance is through impairment of B-cell function and compensatory hyperinsulinemia in predisposed Latinos with insulin resistance and that HCV eradication improves these abnormalities. This study addresses changes in the metabolic parameters over time. In addition, it is hypothesized that moderate alcohol consumption impacts insulin resistance and secretion and 30 patients with or without HCV who drink alcohol moderately will have discontinuation of alcohol use for 6 weeks and have metabolic testing before and after alcohol discontinuation.

ELIGIBILITY:
Inclusion criteria for HCV participants:

* Male or female patients between 18 and 60 years of age
* Body mass index (BMI) > 20 Kg/m2
* Serologic evidence of hepatitis C infection by anti-HCV antibody
* Detectable plasma HCV-RNA
* Compensated liver disease with the following minimum biochemical parameters: prothrombin time < 2 seconds prolonged compared to control and bilirubin < 3 mg/dL
* Willingness to provide informed consent

Inclusion criteria for healthy Latino volunteers (without HCV infection):

-Same inclusion criteria as above except no evidence of HCV infection (anti-HCV antibody negative)

Inclusion criteria for participation in 6-week alcohol abstinence follow-up testing:

-Latinos who are moderate1 alcohol drinkers (1NIAAA definition: female: no more than 3 drinks on any day & no more than 7 drinks per week; male: no more than 4 drinks on any day and no more than 14 drinks per week).

Steady-State Plasma Glucose < 180 mg/dL

Exclusion criteria:

* Hepatitis B or HIV infection
* Subjects with liver disease other than that caused by HCV
* Known history of diabetes, or fasting plasma glucose concentration >126 mg/dl
* Known history of cirrhosis of the liver, as well as individuals with decompensated liver disease such as those with ascites, variceal bleeding, and encephalopathy
* Known history of pancreatitis
* Prior or current treatment for HCV
* Heavy alcohol use (>80 g/d)
* Subjects of lipid lowering agents, steroid/ anabolic therapy
* Significant medical illness that would interfere with the completion of the study

Exclusion criteria for healthy (non HCV) Latino volunteers:

-Same as above, including subjects with HCV infection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Latinos with and without HCV infection
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
insulin resistance | baseline, 6 weeks and 18 months
  steady state plasma glucose level (mg/dL)

SECONDARY OUTCOMES:
Insulin secretion | baseline, 6 weeks and 18 months
  insulin secretion rate area under the curve (pmol/min)

CONTACTS AND LOCATIONS:
Overall Officials: Mandana Khalili, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of california San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Uribe LA, Bacchetti P, Gelman N, Burchard E, Fitch M, Hellerstein M, Khalili M. Impact of Moderate Alcohol Discontinuation on Insulin Action and Secretion in Latinos With and Without Hepatitis C. Alcohol Clin Exp Res. 2018 Mar;42(3):492-499. doi: 10.1111/acer.13576. Epub 2018 Feb 1. PMID 29220547
- [Result] Burman BE, Bacchetti P, Khalili M. Moderate Alcohol Use and Insulin Action in Chronic Hepatitis C Infection. Dig Dis Sci. 2016 Aug;61(8):2417-2425. doi: 10.1007/s10620-016-4119-0. Epub 2016 Mar 23. PMID 27007134
- [Result] Burman BE, Bacchetti P, Ayala CE, Gelman N, Melgar J, Khalili M. Liver inflammation is a risk factor for prediabetes in at-risk latinos with and without hepatitis C infection. Liver Int. 2015 Jan;35(1):101-7. doi: 10.1111/liv.12676. Epub 2014 Sep 20. PMID 25156890
- [Result] Kim RG, Kramer-Feldman J, Bacchetti P, Grimes B, Burchard E, Eng C, Hu D, Hellerstein M, Khalili M. Disentangling the impact of alcohol use and hepatitis C on insulin action in Latino individuals. Alcohol Clin Exp Res. 2022 Jan;46(1):87-99. doi: 10.1111/acer.14743. Epub 2021 Nov 23. PMID 34773280
- [Result] Gonzales CA, Bacchetti P, Khalili M. Impact of gender and menopausal status on metabolic parameters in chronic hepatitis C infection. J Viral Hepat. 2016 Mar;23(3):232-9. doi: 10.1111/jvh.12487. Epub 2015 Nov 10. PMID 26554398
- [Result] Shah SC, Kornak J, Khalili M. Depression is not associated with peripheral insulin resistance in patients with chronic hepatitis C infection. J Viral Hepat. 2015 Mar;22(3):272-80. doi: 10.1111/jvh.12306. Epub 2014 Sep 8. PMID 25196736
- [Result] Mukhtar NA, Bacchetti P, Ayala CE, Melgar J, Christensen S, Maher JJ, Khalili M. Insulin sensitivity and variability in hepatitis C virus infection using direct measurement. Dig Dis Sci. 2013 Apr;58(4):1141-8. doi: 10.1007/s10620-012-2438-3. Epub 2012 Oct 21. PMID 23086116
- [Result] Brandman D, Bacchetti P, Ayala CE, Maher JJ, Khalili M. Impact of insulin resistance on HCV treatment response and impact of HCV treatment on insulin sensitivity using direct measurements of insulin action. Diabetes Care. 2012 May;35(5):1090-4. doi: 10.2337/dc11-1837. Epub 2012 Mar 7. PMID 22399695
- [Result] Mukhtar NA, Ayala C, Maher JJ, Khalili M. Assessment of factors associated with pre-diabetes in HCV infection including direct and dynamic measurements of insulin action. J Viral Hepat. 2012 Jul;19(7):480-7. doi: 10.1111/j.1365-2893.2011.01568.x. Epub 2011 Dec 18. PMID 22676360
- [Result] Lam KD, Bacchetti P, Abbasi F, Ayala CE, Loeb SM, Shah V, Wen MJ, Reaven GM, Maher JJ, Khalili M. Comparison of surrogate and direct measurement of insulin resistance in chronic hepatitis C virus infection: impact of obesity and ethnicity. Hepatology. 2010 Jul;52(1):38-46. doi: 10.1002/hep.23670. PMID 20578127